CLINICAL TRIAL: NCT06634940
Title: International Surveillance of Antimicrobial Resistance in Cirrhosis-Related Infections
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, SEBASTIAN MARCIANO. MD, MsC, Head of Hepatology, Hospital Italiano de Buenos Aires
Other Study IDs: 5821
Record Dates: First submitted 2024-10-06; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cirrhosis; Bacterial Infections; Multidrug Resistance
Keywords: antibiotics; empirical treatment; methicillin-resistant Staphylococcus aureus; extended-spectrum beta-lactamase-producing organisms; Carbapenemase-Producing Enterobacteriaceae; de-escalation; guidelines; empiric antibiotics
MeSH Terms: conditions — Fibrosis; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
What is this study about?

This study tracks antibiotic resistance in patients with cirrhosis who develop bacterial infections. Cirrhosis is a condition where the liver is severely scarred, and people with cirrhosis are at high risk for serious bacterial infections.

Why is this study important?

Bacterial infections are common in patients with cirrhosis, affecting 25-46% of those who are hospitalized. These infections can be life-threatening, with 1 in 4 patients dying from complications. Many of these infections are becoming harder to treat because the bacteria are resistant to antibiotics. Infections caused by resistant bacteria are increasing, which makes finding the right antibiotic quickly even more difficult.

In other regions of the world, guidelines exist to help doctors choose the right antibiotics for cirrhosis patients. However, in Latin America, we don't have specific guidelines for our region, and doctors currently rely on recommendations from the U.S. or Europe. These guidelines may not reflect the local patterns of bacterial infections and resistance we see here.

What is the goal of this study?

The main goal of this study is to create a long-term system to track how bacteria respond to antibiotics in patients with cirrhosis in Latin America. By collecting data from hospitals across different countries, we aim to:

* Identify how many infections are caused by multidrug-resistant bacteria.
* Understand how antibiotics (such as ceftriaxone, vancomycin, and carbapenems) act against these infections.
* Generate reports informing bacterial resistance patterns to help doctors make better patient treatment decisions.

What do we hope to achieve?

We hope the data we collect will help develop guidelines for patients with cirrhosis in Latin America. These guidelines will ensure that doctors use the most effective antibiotics based on real-time data from our region. This should improve patient outcomes and help prevent the spread of resistant bacteria.

DETAILED DESCRIPTION:
Bacterial infections are among the most common complications in patients with cirrhosis, affecting 25-46% of those hospitalized. In two-thirds of cases, these infections are diagnosed during hospitalization, while the remainder develop during the hospital stay. The high mortality rate associated with these infections is significant, with one in four patients succumbing to the complication.

Regarding origin, 30-35% of bacterial infections in patients with cirrhosis are classified as spontaneous, with the rest being non-spontaneous. Spontaneous bacterial peritonitis is the most frequently reported infection specific to patients with cirrhosis and portal hypertension. Other spontaneous infections include spontaneous bacteremia and spontaneous bacterial empyema.

A significant factor influencing patient outcomes in bacterial infections is the rapid initiation of appropriate empirical antibiotic therapy. It is generally recommended that empirical treatment covers 80% of expected bacteria in stable patients and 90% in critically ill patients. However, this goal is increasingly challenging due to shifting epidemiology, with a rise in Gram-positive organisms and a growing incidence of multidrug resistance. Recent studies have shown that 34% of infections in patients with cirrhosis are caused by multidrug-resistant microorganisms, which are linked to poorer outcomes, complicating patient management, and increasing healthcare costs.

Although guidelines for empirical antibiotic treatment exist in other regions, none have been developed for Latin America. As a result, clinicians often rely on recommendations from the United States or Europe, which may not accurately reflect the epidemiology in this region.

GENERAL OBJECTIVES

1. To establish and sustain a surveillance system to monitor the antibiotic susceptibility patterns of microorganisms responsible for infections in patients with cirrhosis.
2. To produce periodic reports on evolving resistance patterns of microorganisms involved in infections in patients with cirrhosis.

EXPECTED OUTCOMES

This project aligns with global strategies to address the rise in infections caused by multidrug-resistant microorganisms. By applying a research methodology based on international standards, the study aims to ensure the collection of high-quality data that can lead to actionable outcomes.

Our research team initiated this project in 2020 to create a continuous surveillance program for bacterial infections in cirrhosis patients within our region. The goal is to collect and share real-time data on antibiotic susceptibility patterns.

We expect to generate results that will enable the production of detailed reports on the susceptibility patterns of bacterial infections in patients with cirrhosis at different levels. This will provide the necessary information to develop region-specific guidelines for the appropriate use of empirical antibiotics in this population. Additionally, periodic updates will reflect ongoing epidemiological changes.

---

This structure improves the flow and maintains a scientific tone. Let me know if further revisions are needed!

ELIGIBILITY:
Inclusion Criteria:

* Episodes of culture-confirmed bacterial infections
* Patients diagnosed with cirrhosis
* Infections diagnosed either at the time of hospital admission or during hospitalization

Exclusion Criteria:

* History of solid organ or hematopoietic stem cell transplantation
* Declined to participate in the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients in Latin American countries
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of multidrug-resistant organisms | 1 week
  Estimated by using the total number of bacterial infection episodes involving at least one multidrug-resistant organism as the numerator and the total number of bacterial infection episodes as the denominator.
Proportion of extensively drug-resistant microorganisms | 1 week
  Estimated by using the total number of bacterial infection episodes involving at least one extensively drug-resistant microorganism as the numerator and the total number of bacterial infection episodes as the denominator.
Proportion of pan drug-resistant microorganisms | 1 week
  Estimated by using the total number of bacterial infection episodes involving at least one pan drug-resistant microorganism as the numerator and the total number of bacterial infection episodes as the denominator.

SECONDARY OUTCOMES:
Proportion of episodes on infection susceptible to quinolones | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to quinolones as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to quinolones for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to nitrofurantoin | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to nitrofurantoin as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to nitrofurantoin for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to Trimethoprim-Sulfamethoxazole | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to Trimethoprim-Sulfamethoxazole as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to Trimethoprim-Sulfamethoxazole for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to ceftriaxone | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to ceftriaxone as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to ceftriaxone for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to ceftazidime | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to ceftazidime as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to ceftazidime for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to cefepime | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to cefepime as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to cefepime for the episode to be considered susceptible
Proportion of episodes of infection susceptible to aminoglycosides | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to aminoglycosides as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to aminoglycosides for the episode to be considered susceptible
Proportion of episodes of infection susceptible to piperacillin-tazobactam | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to piperacillin-tazobactam as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to piperacillin-tazobactam for the episode to be considered susceptible
Proportion of episodes of infection susceptible to ertapenem | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to ertapenem as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to ertapenem for the episode to be considered susceptible
Proportion of episodes of infection susceptible to meropenem/imipenem | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to meropenem or imipenem as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to meropenem or imipenem for the episode to be considered susceptible
Proportion of episodes of infection susceptible to colistin: | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to colistin as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to colistin for the episode to be considered susceptible
Proportion of episodes of infection susceptible to ceftazidime-avibactam | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to ceftazidime-avibactam as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to ceftazidime-avibactam for the episode to be considered susceptible
Proportion of episodes of infection susceptible to ceftolozane-tazobactam | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to ceftolozane-tazobactam as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to ceftolozane-tazobactam for the episode to be considered susceptible
Proportion of episodes of infection susceptible to piperacillin-tazobactam plus vancomycin | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to piperacillin-tazobactam or vancomycin as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to at least one of the antibiotics for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to carbapenem plus vancomycin | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to both carbapenem and vancomycin as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to both antibiotics for the episode to be considered susceptible
Proportion of episodes of infection susceptible to carbapenem plus linezolid | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to carbapenems or linezolid as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to at least one of the antibiotics for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to carbapenem + linezolid | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to either carbapenem or linezolid as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to at least one of the antibiotics for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to aminoglycoside + colistin | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to either aminoglycoside or colistin as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to at least one of the antibiotics for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to ceftazidime-avibactam + aztreonam | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to either ceftazidime-avibactam or aztreonam as the numerator and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to at least one of the antibiotics for the episode to be considered susceptible.
Proportion of episodes of infection susceptible to ceftazidime-avibactam + vancomycin | 1 week
  Estimated by using the total number of bacterial infection episodes involving microorganisms with in vitro susceptibility to either ceftazidime-avibactam or vancomycin as the numerator, and the total number of bacterial infection episodes as the denominator. For episodes involving more than one organism, all organisms must be susceptible to at least one of the antibiotics for the episode to be considered susceptible

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
I am willing to share individual participant data based on the proposal, the project's relevance and importance, and ensuring data security
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: form October 2024 to October 2030